CLINICAL TRIAL: NCT02937987
Title: Dietary Intake, Eating Behavior, Physical Activity Level and Their Relationships With Glycemic and Weight Control in Hong Kong Chinese Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lorena Tsui Fun Cheung, PhD student in medical science, Chinese University of Hong Kong
Other Study IDs: Lifestyle-001
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes Mellitus in Obese

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group 1: non-obese type 2 DM
- Group 2: obese type 2 DM

SUMMARY:
The objective of this study is to describe and examine the dietary intake, eating behavior and physical activity level of a cohort of Hong Kong Chinese with T2DM and their association with weight and glycemic control at baseline and 1 year follow-up. The investigators hypothesize that Hong Kong Chinese T2DM patients with unhealthy dietary intake and pattern and low physical activity level are associated with poorer glycemic and weight control, and there will be no improvement with weight and glycemic control under usual care after 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of Chinese ethnicity
2. Diagnosis of T2DM
3. Able to read Chinese and give informed written consents

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. End-stage renal failure requiring dialysis or chronic kidney disease (CKD) stage 4 or above
3. Malignancy diagnosed within 3 years
4. Pregnancy or lactation
5. Any medical illness or condition as judged by the investigators as ineligible to participate the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hong Kong Chinese T2DM patients referred to the Prince of Wales Hospital (PWH) diabetes centre
Sampling Method: Non-Probability Sample
Enrollment: 211 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c | 1 year
Change of Weight | 1 year